CLINICAL TRIAL: NCT04022902
Title: The Experience of Patients and Family Caregivers in Managing Pneumoconiosis in the Family Context: An Exploratory Qualitative Study
Brief Title: The Experience of Patients and Family Caregivers in Managing Pneumoconiosis in the Family Context
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Li Wai Chi Polly, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: PCFB2018
Record Dates: First submitted 2019-07-12; First posted 2019-07-17 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Pneumoconiosis
Keywords: Pneumoconiosis; Self-care; Care-giving
MeSH Terms: conditions — Pneumoconiosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This is an exploratory qualitative study to understand the needs of patients with pneumoconiosis, and the care-giving experience of their family caregivers.
  Other Names: Qualitative study

SUMMARY:
This is an exploratory qualitative study to understand the needs of patients with pneumoconiosis, and the care-giving experience of their family caregivers. Patients with a confirmed diagnosis of pneumoconiosis for at least 1 year and had registered with the Pneumoconiosis Compensation Fund Board in Hong Kong to receive compensation will be eligible to join this study. The respective family caregivers of these patients, who are 21 years of age or older, assuming the role as the primary caregivers of a pneumoconiosis patient who have registered with the Pneumoconiosis Compensation Fund Board will be invited to join. The nurse will carry out an individual in-depth qualitative interview at patient's home. The nurse will also conduct a home environment assessment. After obtaining the written consent, an interview guide with a list of open-ended questions will be used to elicit the illness experience and self-care needs of the pneumoconiosis patients and the caregiving experience of their family caregivers.

DETAILED DESCRIPTION:
Pneumoconiosis is a fibrotic pulmonary disease resulting from workplace exposure to hazardous dusts containing free silica or asbestos, which causes irreversible progressive respiratory impairment among the sufferers. These patients may experience disabling symptoms (e.g. progressive severe dyspnea, chronic and uncontrolled cough, sputum production, fatigue, activity intolerance, decreased mobility and sleep disturbance) despite optimal medical treatment. Pneumoconiosis is considered as a chronic, progressive and incurable disease which requires long-term comprehensive rehabilitation services and support. Effective disease management relies on engaging patients in long-term comprehensive rehabilitation. The overall aim of this study is to explore the illness experience and needs of patients with pneumoconiosis, and the caregiving experience of their respective family caregivers through home visits. The findings will provide important insight into the development of an effective and tailor-made support program for patients with pneumoconiosis in Hong Kong.

This is an exploratory qualitative study to understand the needs of patients with pneumoconiosis, and the care-giving experience of their family caregivers. Patients with a confirmed diagnosis of pneumoconiosis for at least 1 year and had registered with the Pneumoconiosis Compensation Fund Board in Hong Kong to receive compensation will be eligible to join this study. The respective family caregivers of these patients, who are 21 years of age or older, assuming the role as the primary caregivers of a pneumoconiosis patient who have registered with the Pneumoconiosis Compensation Fund Board will be invited to join. The nurse will carry out an individual in-depth qualitative interview at patient's home. The nurse will also conduct a home environment assessment, as the home environment plays an important role in promoting or restricting performance of everyday tasks of people with disabling chronic diseases and their caregivers. The interviews will be conducted with the patients and the caregivers separately, so they can talk openly and confidentiality is guaranteed. Prior to commencement of the data collection, the nurse will provide an information sheet to solicit participants' understanding about the nature of the study, their rights and confidentiality issues. After obtaining the written consent, an interview guide with a list of open-ended questions will be used to elicit the illness experience and self-care needs of the pneumoconiosis patients and the caregiving experience of their family caregivers. All the interviews will be audio-taped after obtaining the permission from the participants.

This study aims to explore the illness experience and needs of patients with pneumoconiosis and the care-giving experience of their caregivers. Specifically, the objectives of this study are as follow:

* To understand the self-care behaviors and illness experience of patients with pneumoconiosis
* To explore the needs of patients with pneumoconiosis when managing the disease at home and in the community
* To understand the caregiving experience of the family caregivers of patients with pneumoconiosis
* To explore the caregivers' needs when taking care of patients with pneumoconiosis
* To explore how disease management and caregiving take place in patients' home environment and to identify the environment-related facilitators and barriers for managing pneumoconiosis.

After the interview, the nurse will also conduct a home environment assessment with a standard environmental checklist to evaluate the home for safety, modification needs and ease of mobility. Such assessment would provide valuable information to inform the needs of pneumoconiosis patients and their caregivers when they participate community-based and home-based rehabilitative activities. The assessment includes the environment outside and within patients' home environment, such as any difficulties in accessing the entrance of the building (e.g. barrier-free entryway, no elevator for one or more floor), the use of equipment or adaptations in the home to aid in daily activities, such as rails and commodes. The commonly seen home environmental hazards will also be assessed, such as the exposure to second-hand smoking, the use of nonskid mats in bathroom, grab bars in the shower or tub, spacing and entryway in the bathroom and bedroom. Each of the item will be assessed to solicit a 'no problem observed' or 'problem observed'.

The audio-taped qualitative data will be transcribed verbatim by the research nurse. Content analysis will be adopted for the data analysis. In particular, the qualitative data will be analyzed to seek a better understanding of what and how the patients and the caregivers can be supported in their disease self-care and caregiving trajectory. The emerged themes from the qualitative data will be used to optimize the patient support program in the subsequent quantitative phase of the study. The home environment assessment data will be summarized by appropriate numbers and percentages.

ELIGIBILITY:
Inclusion Criteria:

For Patients:

* a confirmed diagnosis of pneumoconiosis for at least 1 year
* had registered with the Pneumoconiosis Compensation Fund Board in Hong Kong to receive compensation

For the respective family caregivers:

* 21 years of age or older
* assuming the role as the primary caregivers of a pneumoconiosis patient who have registered with the Pneumoconiosis Compensation Fund Board

Exclusion Criteria:

* Those patients or family caregivers with impaired communication ability or impaired cognitive function [as indicated by the Abbreviated Mental Test (AMT) score ≤ 6/10] in preventing them to participate in the research activities will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pneumoconiosis patient who have registered with the Pneumoconiosis Compensation Fund Board. Their primary caregivers will be invited to join as well.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Experience of self-management of pneumoconiosis | 60 minutes
  Evaluation from the patients' point of view on how they self-manage pneumoconiosis in the community and what are their unmet needs, semi-structured qualitative interviews with pneumoconiosis patients will be conducted.
Care-giving experience of family caregivers of pneumoconiosis | 60 minutes
  Evaluation from the family caregivers' point of view on their care-giving experience of patients with pneumoconiosis and their needs when taking care of their care recipients. semi-structured qualitative interviews with the family caregivers of pneumoconiosis patients will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Polly Li, Prof, Principal Investigator — The Nethersole School of Nursing
Locations (1):
- Pneumoconiosis Compensation Fund Board, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li PWC, Yu DSF, Tam SYS. The experience of patients and family caregivers in managing pneumoconiosis in the family context: A study protocol. J Adv Nurs. 2019 Dec;75(12):3805-3811. doi: 10.1111/jan.14203. Epub 2019 Oct 2. PMID 31576609